CLINICAL TRIAL: NCT00924001
Title: Phase I/II Study Using a Non-Myeloablative Lymphocyte Depleting Regimen of Chemotherapy Followed by Infusion of Allogeneic Tumor-Reactive Lymphocyte Cell Line DMF5 in Metastatic Melanoma
Brief Title: Chemotherapy Followed by Infusion of DMF5 Cells to Treat Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: study was stopped due to low accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Steven A. Rosenberg, M.D./National Cancer Institute, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070210; 07-C-0210; NCT00537069 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-06-07 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Melanoma; Malignant Melanoma; Melanoma, Experimental
Keywords: Clinical Response; Immunotherapy; Cancer; Cytokines; Adoptive Cell Therapy; Melanoma; Metastatic Melanoma
MeSH Terms: conditions — Melanoma; Melanoma, Experimental; Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metastatic Melanoma (Experimental): Melanoma that has invaded deep into the skin, lymph nodes, or other parts of the body.
  Interventions: Drug: DMF5 Melanoma Reactive TIL; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: Aldesleukin

INTERVENTIONS:
Drug: DMF5 Melanoma Reactive TIL — given intravenously over 20-30 minutes (between 1 x 10^9 and 1 x 10^11 lymphocytes) after expansion in interleukin-2 and OKT-3
Drug: Cyclophosphamide — 60 mg/kg/day x 2 days intravenously
  Other Names: Cytoxan; Endoxan; Neosar; Procytox; Revimmune
Drug: Fludarabine — 25 mg/m^2/day intravenously x 5 days
  Other Names: Fludara
Drug: Aldesleukin — 720,000 IU/kg/dose intravenously every 8 hours for up to 15 doses
  Other Names: Proleukin

SUMMARY:
Background:

* This study will use cells called DMF5 to treat patients with metastatic melanoma (melanoma that has spread beyond the primary tumor site).
* The DMF5 cells were first obtained from a tumor of a patient with melanoma with HLA-A201 tissue type. The tumor cells were grown in the laboratory, and when the laboratory-grown cells were given back to the patient, the patient's tumors shrank dramatically. In laboratory tests, DMF5 cells were also shown to shrink mouse melanoma tumors.

Objectives:

-To determine whether preparatory chemotherapy followed by infusion of DMF5 cells is a safe and effective for shrinking melanoma tumors.

Eligibility:

-Patients with metastatic melanoma and tissue type HLA-A201 who are 18 years of age or older.

Design:

* Patients have a preparatory regimen of chemotherapy with cyclophosphamide and fludarabine followed by infusion of DMF5 cells and then high-dose interleukin. The chemotherapy, interleukin and cells are given intravenously (through a vein).
* Patients have frequent blood tests to look for the side effects and response to treatment.
* Patients may be asked to have a tumor biopsy (surgical removal of a small piece of tumor tissue) to examine the effects of treatment on the immune cells in the tumor.
* Patients have a physical examination, computed tomography (CT) of the chest, abdomen and pelvis and laboratory tests 4 to 6 weeks after treatment and then monthly to evaluate the tumor.
* The first group of patients participates in the Phase I portion of the study, called the dose escalation phase. This phase will determine the highest safe dose of DMF5 cells. There will be three dose levels of DMF5 cells, with the first patients enrolled getting the smallest dose and then increasing the dose when the preceding level has been shown to be safe.
* Patients in the Phase II portion of the study receive DMF5 cells at the highest dose found to be safe in Phase I, to test the effectiveness of the treatment.

DETAILED DESCRIPTION:
Background:

In previous trials in the Surgery Branch, a 51 percent objective response rate has been observed in heavily pre-treated patients with metastatic melanoma undergoing adoptive cell transfer therapy utilizing a non-myeloablative preparative regimen followed by administration of autologous tumor-reactive lymphocytes and subsequent treatment with high-dose aldesleukin.

However, in patients with metastatic melanoma undergoing metastasectomy, recovery of adequate numbers of tumor specific T lymphocytes from surgical specimens is possible in approximately half of all patients, thus limiting the application of adoptive cell transfer therapy.

Murine models performed in the Surgery Branch have demonstrated solid tumor regression in mice treated with allogeneic tumor specific T cells combined with a preinfusion lymphodepleting regimen.

We have identified a tumor specific lymphocyte cell line (DMF5) used previously in an autologous adoptive cell transfer protocol that was associated with an objective clinical response in that patient.

In subsequent preclinical testing of this lymphocyte population, we have demonstrated high specificity against HLA-A 0201 positive melanoma cell lines as well as the common shared melanocyte differentiation antigen MART-1:27-35. We have expanded this lymphocyte population to provide up to 30 individual allogeneic cell transfers to HLAA 0201 positive patients with metastatic melanoma.

In this trial we want to test our hypothesis that objective tumor regression can be achieved with the DMF5 allogeneic T-cell product using a non-myeloablative regimen followed by cell transfer and high-dose aldesleukin.

It should be emphasized that this protocol is designed to test whether highly melanoma reactive allogeneic lymphocytes can mediate cancer regression. The DMF5 cell line is a limited reagent only available for the treatment of up to 30 patients. However, if this treatment results in cancer regression, it will represent an important step in our development of an allogeneic T-cell receptor engineered universal effector cell line for the treatment of patients with cancer.

Objectives:

To evaluate the safety of the administration of the DMF5 allogeneic T-cell product in patients receiving the non- myeloablative conditioning regimen, and aldesleukin.

To determine whether this allogeneic tumor-specific lymphocyte cell line, hereafter referred to as DMF5, infused in conjunction with the administration of high-dose aldesleukin may result in objective clinical tumor regression in eligible HLA-A 0201 positive patients with metastatic melanoma receiving a non-myeloablative lymphoid depleting preparative regimen.

To determine the in vivo survival of the infused cells following the non-myeloablative regimen, via analysis of the sequence of the variable region of the T cell receptor or flow cytometry (FACS).

Eligibility:

Patients with metastatic melanoma who are greater than or equal to 18 years of age, HLA-A 0201 positive, do not have suitable autologous tumor reactive TIL cells available, and are able to tolerate high-dose aldesleukin.

Design:

Patients will receive a non-myeloablative lymphocyte depleting preparative regiment consisting of cyclophosphamide (60 mg/kg/day times 2 days intravenous (IV)) and fludarabine (25 mg/m2/day IV times 5 days).

Patients will receive intravenous adoptive transfer of the tumor reactive lymphocyte cell line DMF5 (after its expansion in interleukin-2 and OKT3) followed by high-dose intravenous (IV) aldesleukin (720,000 IU/kg/dose every 8 hours for up to 15 doses).

Patients will undergo complete evaluation of tumor with physical examination, CT of the chest, abdomen, and pelvis and clinical laboratory evaluation four to six weeks after treatment and then monthly for approximately 3 to 4 months or until off study criteria are met. The study will be conducted using a Phase I/II optimal design. The protocol will proceed in a phase 1 dose escalation design, with three cohorts. Should a single patient experience a dose limiting toxicity at a particular dose level, three more patients would be treated at that dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level with 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose prior to starting the phase II portion. If a dose limiting toxicity occurs in the first cohort, that cohort will be expanded to 6 patients. If 2 DLTs are encountered in this cohort, the study will be terminated.

Once the MTD has been determined, the study then would proceed to the phase II portion, and initially, 9 total patients will be administered the therapy at the maximum tolerated dose. The plan will utilize a Simon two-stage optimal phase II design. If 0 of the 9 patients experiences a clinical response, then no further patients will be enrolled but if 1 or more of the first 9 evaluable patients enrolled have a clinical response, then accrual will continue until a total of 30 evaluable patients have been enrolled.

This design has the ability to distinguish a 5% response rate (p0=0.05) from a 25% response rate (p1=0.25), with 10% probability of falsely "accepting" the DMF5 cell therapy approach (alpha=0.10), and 10% probability of incorrectly discarding this strategy as if it were unacceptably poor (beta=0.10). This design also has 63% probability of stopping early (at 9 patients) if the true response rate is 5%.

ELIGIBILITY:
-INCLUSION CRITERIA:

1. Measurable metastatic melanoma that is refractory to standard treatment including high dose aldesleukin.
2. Unsuitable autologous cells for Institutional Review Board (IRB) approved Surgery Branch adoptive cell therapy studies.
3. Greater than or equal to 18 years of age.
4. Life expectancy of greater than three months.
5. Willing to sign a durable power of attorney.
6. Able to understand and sign the Informed Consent Document.
7. Human leukocyte antigen A (HLA-A) 0201 positive.
8. Willing to practice birth control during treatment and for four months after receiving the preparative regimen.
9. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
10. Hematology:

    * Absolute neutrophil count greater than 1000/mm^3 without support of filgrastim.
    * WBC greater than 3000/mm^3.
    * Hemoglobin greater than 8.0 g/dl.
    * Platelet count greater than 100,000/mm^3.
11. Serology:

    * Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune - competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
    * Seronegative for hepatitis B antigen and hepatitis C antibody unless antigen negative.
12. Chemistry:

    * Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less than three times the upper limit of normal.
    * Serum creatinine less than or equal to 1.6 mg/dl.
    * Total bilirubin less than or equal to 2.0 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
13. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).
14. Six weeks must have elapsed since prior Ipilimumab (MDX-010) therapy to allow antibody levels to decline.
15. Patients who have previously received MDX-010 must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Opportunistic infections (The experimental treatment being evaluated in his protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities.)
5. Symptomatic central nervous system (CNS) lesions (Patients maybe eligible after treatment of their symptomatic lesions.)
6. Systemic steroid therapy.
7. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
8. History of coronary revascularization or ischemic symptoms.
9. Patients with a prolonged (greater than 20 pk/yrs) history of cigarette smoking or symptoms of respiratory dysfunction with pulmonary function tests (PFT's) indicating an forced expiratory volume (FEV1) less than 60 percent predicted for age.
10. Patients with a history of clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, heart block or greater than or equal to age 60 with an left ventricular ejection fraction (LVEF) of less than 45 percent on cardiac evaluation (echocardiogram, multi-gated acquisition scan (MUGA), etc.) will be excluded.
11. Positive allo-specific reactivity of the DMF5 cells to the patient's peripheral blood mononuclear cells (PBMC).
12. Documented penicillin allergy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2007-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rosenberg, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Mills CD, North RJ. Expression of passively transferred immunity against an established tumor depends on generation of cytolytic T cells in recipient. Inhibition by suppressor T cells. J Exp Med. 1983 May 1;157(5):1448-60. doi: 10.1084/jem.157.5.1448. PMID 6189937
- [Background] Fernandez-Cruz E, Woda BA, Feldman JD. Elimination of syngeneic sarcomas in rats by a subset of T lymphocytes. J Exp Med. 1980 Oct 1;152(4):823-41. doi: 10.1084/jem.152.4.823. PMID 6968337
- [Background] Greenberg PD, Kern DE, Cheever MA. Therapy of disseminated murine leukemia with cyclophosphamide and immune Lyt-1+,2- T cells. Tumor eradication does not require participation of cytotoxic T cells. J Exp Med. 1985 May 1;161(5):1122-34. doi: 10.1084/jem.161.5.1122. PMID 3921652

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One participant was enrolled to this study.
Period: Overall Study
Arm/Group | Metastatic Melanoma
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 32.0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With an Objective Clinical Tumor Regression Response According to RECIST Criteria
Description: Response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST). Complete response (CR) is the disappearance of all target lesions, partial response (PR) is at least a 30% decrease in the target lesions, progression (PD) is at least a 20% increase in the target lesions or appearance of one or more new lesions, and stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Time Frame: 44 days
Measure: Number; unit: Participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 1
Participants | 0

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here are the number of participants with adverse events. For a detailed list of adverse events see the adverse event module.
Time Frame: 44 days
Measure: Number; unit: Participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 1
Participants | 1

3. Secondary Outcome: Number of Participiants With In-vivo Survival of Infused Cells
Description: In-vivo survival of infused cells is determined by analysis of the sequence of the variable region of the T cell receptor or flow cytometry (FACS).
Time Frame: 44 days
Measure: Number; unit: Participants
Arm/Group | Metastatic Melanoma
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 44 days
Arm/Group | Metastatic Melanoma
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metastatic Melanoma (N=1)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (1)
Leukocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Lymphocyte count decreased (Blood and lymphatic system disorders) | 1 (1)
Neutrophil count decreased (Blood and lymphatic system disorders) | 1 (1)
Platelet cout decreased (Blood and lymphatic system disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (2)
Oral pain (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No